CLINICAL TRIAL: NCT05781737
Title: Inflammatory Bowel Disease and Atherosclerosis Development
Status: Active, not recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, Professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 22-22
Record Dates: First submitted 2023-01-16; First posted 2023-03-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Diseases; Cardiovascular Diseases; Inflammation; Arterial Stiffness
MeSH Terms: conditions — Inflammatory Bowel Diseases; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ulcerative colitis
- Crohn disease
- Control group

SUMMARY:
The study will show the influence of inflammatory bowel disease on the risk of development of atherosclerosis

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Other conditions affecting the prognosis
* Psychiatric disorders affecting the participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with ulcerative colitis, 50 patients with Crohn disease, 50 patients without inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Intima-media thickness | 1 year
  Intima-media thickness
Pulse wave velocity | 1 year
  Pulse wave velocity

SECONDARY OUTCOMES:
All cause mortality | 1 year
Cardiovascular mortality | 1 year
Hospitalisation due to cardiovascular disease | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital #1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Isaikina M.A., Isaev G.O., Pyatigorets E.S., Yurazh M.A., Mironova O.I. Ulcerative colitis and cardiovascular disease. Case report. Systemic Hypertension. 2022;19(4):53-57. (In Russ.) — https://doi.org/10.38109/2075-082X-2022-4-53-57